CLINICAL TRIAL: NCT07013331
Title: A PET-MRI Study of Serotoninergic Brainstem Pathway in Patients With Dravet Syndrome
Acronym: DRAPETONINE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 69HCL24_1231
Record Dates: First submitted 2025-04-25; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy; Dravet Syndrome; Drug Resistant Epilepsy; Healthy Controls
Keywords: epilepsy; Dravet syndrome; drug-resistant focal epilepsy; serotonin; PET-MRI; MPPF; SUDEP
MeSH Terms: conditions — Epilepsy; Epilepsies, Myoclonic; Drug Resistant Epilepsy; Sudden Unexpected Death in Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with Dravet syndrome (Experimental): Adult patients with Dravet syndrome (> 18 and < 60 years). Diagnosis of Dravet syndrome will be confirmed based on medical history, type of seizures, EEG data and results of genetic testing. Ten DS patients will be recruited and will be passed the PET-IRM with injection of the tracer [18F]MPPF.
  Interventions: Other: [18F]MPPF PET-MRI
- Patients with drug-resistant focal epilepsy (Experimental): Adult patients (> 18 years) with drug-resistant focal epilepsy, as defined by the ILAE, and whom presurgical evaluation is considered. Ten patients will be recruited and will be passed the PET-IRM with injection of the tracer [18F]MPPF.
  Interventions: Other: [18F]MPPF PET-MRI
- Adult healthy controls (> 18 years) (Experimental): Ten healthy controls will be recruited and will be passed the PET-IRM with injection of the tracer [18F]MPPF. Participants must be of legal age.
  Interventions: Other: [18F]MPPF PET-MRI

INTERVENTIONS:
Other: [18F]MPPF PET-MRI — Patients will be seen during an first inclusion visit during which a review of eligibility criteria, medical history and a clinical examination will be done. Participants will be scheduled for a PET-MRI scan within 2 to 8 weeks. For all women of childbearing age a urine pregnancy test will be performed before the PET-MRI.
  Anatomical MR imaging will be first acquired for anatomical co-registration and morphometry analyses (Neuromelanin sensitive images and 3D anatomical T1-weighted covering the whole brain volume with 1mm3 cubic voxels) After i.v. injection of a bolus of 180 MBq ± 10%, with a maximum of 198 MBq MBq, of [18F]-MPPF, a dynamic emission scan consisting of 35 frames of increasing duration (20s to 5min) will be acquired over 90-min post-injection

SUMMARY:
Dravet Syndrome (DS) is a severe neurodevelopmental disease, which is predominantly caused by mutations of SCN1A, the gene coding for Nav1.1 voltage-gated sodium channels. DS is characterized by infancy onset, severe cognitive deficit and drug-resistant seizures, including several generalized convulsive seizures per day and frequent status epilepticus, often triggered by fever or hyperthermia. Among the causes of premature deaths in patients with epilepsy, sudden and unexpected death in epilepsy (SUDEP) represents a major cause. SUDEP is a non-traumatic and non-drowning death in patients with epilepsy, unrelated to a documented status epilepticus. The risk of SUDEP is particularly high in patients suffering from DS, reaching about 9/1000-person-year, as compared to about 1/1000-person-year in people with epilepsy including all disease types. The main clinical risk factor of SUDEP is the frequency of convulsive seizures. Beyond improving seizure control, which we showed to mitigate the SUDEP risk, more specific preventive treatment strategies are still lacking.

Experimental and clinical data suggest that most SUDEP cases result from postictal brainstem dysfunction, including central respiratory arrest There is a body of evidence suggesting involvement of serotonin (5HT) dysfunction both in the pathogenesis of epilepsy in DS and in seizure-related respiratory dysfunction. Serotonin indeed plays a key role in the regulation of respiration. Population firing of serotoninergic neurons in the medullary raphe is significantly decreased during the ictal and post-ictal periods, in association with decreased breathing and heart rate during and after seizures. Most importantly, post-mortem data in patients, including DS, showed alteration of neuronal populations in the medulla in SUDEP cases with evidence for greater reduction in neuromodulatory neuropeptidergic and monoaminergic, including serotoninergic, systems.

SUDEP in DS might therefore be the result of a seizure-induced fatal apnea in a patient who has developed epilepsy-related vulnerability to central respiratory dysfunction favored by 5HT dysfunction. However, several issues remain to be addressed to identify detailed mechanisms and effective therapies. Among them, a key issue is the exact relation between the alterations of the 5HT pathway observed in DS and epilepsy-related respiratory dysfunction

In the present study, the hypothesis is that adult patients with DS might demonstrate specific alterations of the 5HT pathway within the brainstem as assessed by PET imaging. The DRAPETOTINE study will thus focus on imaging 5HT brainstem pathway with PET and MRI in patients with DS to assess if abnormalities can be observed and through comparison with data collected in patients drug-resistant focal epilepsy whether these abnormalities are DS specficic or reflect the consequence on brainstem 5HT pathway of refractory seizures.

This study will involve 20 adult patients, including 10 adults with established diagnosis of Dravet Syndrome and 10 patients with drug-resistant focal epilepsy. Ten healthy adults will also be included. Participants will be recruited over a period of 18 months and the duration of participation for each participant will be 2 weeks to 8 weeks

ELIGIBILITY:
Patients with DS

* Inclusion criteria

  * Adult patients (≥ 18 but < 60 years) with established diagnosis of Dravet Syndrome
  * Adults protected by a guardianship or curatorship
  * Diagnosis of Dravet syndrome will be confirmed based on medical history, type of seizures, EEG data and results of genetic testing
  * No restriction related to the seizure frequency
  * Patient (or patient's legal representative) who gave its written informed consent to participate to the study
  * Patient and/or Legal representative understanding and speaking national language
  * Absence of known current pregnancy and breastfeeding
  * Patient affiliated to the French national health care system
* Exclusion criteria

  * Subject in exclusion period of another study
  * MRI contra-indication (presence of metallic elements)
  * Presence of Vagal Nerve Stimulation
  * Claustrophobia
  * Patients unable to maintain a minimul level of immobility during the imaging acquisition

Patients with drug-resistant focal epilepsy

* Inclusion criteria

  * Adult patient (≥ 18 years) suffering from drug-resistant focal epilepsy according to ILAE classification
  * Patients in whom presurgical evaluation is considered
  * Patient who gave her/his written informed consent to participate to the study
  * No restriction related to the seizure frequency
  * Absence of known current pregnancy and breastfeeding
  * Patient affiliated to French health care system
* Exclusion criteria

  * Subject in exclusion period of another study
  * Adults protected by a guardianship or curatorship
  * MRI contra-indication (presence of metallic elements)
  * Presence of Vagal Nerve Stimulation
  * Claustrophobia
  * Ongoing serotoninergic treatment, including selective serotonin reuptake inhibitor

Healthy controls

* Inclusion criteria

  * Adult (≥ 18 years)
  * Without history of neurological disorders and/or psychiatric disorders, and/or general medical disorders
  * Subject who gave her/his written informed consent to participate to the study
  * Subject affiliated to the French health care system
  * Absence of known current pregnancy and breastfeeding
* Exclusion criteria

  * Age < 18 years
  * Presence of the symptoms of anxiety and/or depression as defined by a score ≥ 11 at the French version of the Hospital Anxiety and Depression Scale (HADS)
  * Ongoing treatment with selective serotonin reuptake inhibitor
  * MRI contra-indication (presence of metallic elements)
  * Claustrophobia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the brainstem BPND of [18F]-MPPF across patients groups (DS and focal epilepsy) | Emission will be acquired over 90 minutes post-injection
  Dynamic PET images will be modelled using a simplified reference tissue model to estimate non-displaceable binding potential (BPND) values in each voxel with reference to the cerebellar white matter excluding the vermis.

SECONDARY OUTCOMES:
Relation between the brainstem BPND of [18F]-MPPF and the total duration of central sleep apneas during total sleep time over a 24-hour period in patients with DS | at Visit 2 (week 2)
  The total duration of central sleep apnea has been preferred to the total number of episodes of central sleep apnea as primary endpoint in order to take into account both the occurrence rate and the severity of episodes. To take into account the variability of the total sleep time across patients, the total duration of central sleep apneas will be expressed as the percentage of the total sleep time for each patient. Sleep apneas can classified as obstructive, central or both central sleep apnea, Apnea will be defined as a decrease in peak nasal pressure of >90% of baseline, lasting at least 10 s. Hypopnea was defined as a decrease of >30% of the baseline nasal pressure, lasting at least 10 s and associated with ≥4% drop in SpO2. Central apnea will be defined by cessation > 10 seconds of airflow with simultaneous cessation of respiratory effort. The respiratory events are scored in clinical routine according to the 2007 American Academy of Sleep Medicine guidelines.
Comparing brainstem volume of patients with DS with the one of patients with drug-resistant focal epilepsy | at Visit 2 (week 2)
  Comparing VBM on the brainstem parcels of patients with DS with the one of patients with drug-resistant focal epilepsy
Relation in DS between brainstem volumes and the total duration of central sleep apneas during total sleep time over a 24-hour period | at Visit 2 (week 2)
Signal-noise radioactivity ratio of 5-HT1A receptors binding in healthy subjects | at Visit 2 (week 2)
  Comparing the signal-noise radioactivity ratio of 5-HT1A receptors binding in healthy subjects with the one observed with the old PET camera used to develop the CERMEP normative database of 5-HT1A receptors binding in adults

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Neurologique Pierre Wertheimer, Bron, Rhone, France

IPD SHARING:
Plan to Share IPD: No